CLINICAL TRIAL: NCT04540029
Title: Measuring Outcomes of Maternal COVID-19-related Prenatal Exposure
Acronym: MOM-COPE
Status: Completed | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MOM-COPE
Record Dates: First submitted 2020-09-02; First posted 2020-09-07 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Prenatal Stress
Keywords: COVID-19; Epigenetics; Prenatal stress; Stress regulation; Maternal sensitivity; Pandemics; Serotonin transporter; Glucocorticoid receptor; Oxytocin receptor; Brain-derived neutropic factor
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Exposed Pregnancy (CEP): Women who were pregnant and delivered during the outbreak of COVID-19 pandemic in Italy, and their infants.
  Interventions: Other: Maternal stress

INTERVENTIONS:
Other: Maternal stress — Prenatal COVID-19-related stress retrospectively self-reported by mothers after delivery.

SUMMARY:
The rapidly spreading coronavirus Covid-19 pandemic is a major concern worldwide and Italy is at the forefront of this emergency. At the present moment, the effects on the offspring of Covid-19 disease in pregnant women and/or the indirect effect of COVID-19-related prenatal maternal stress are poorly understood. Epigenetic mechanisms - and especially DNA methylation - are involved in the embedding of prenatal exposures to large-scale disasters into the epigenome and phenotypic outcomes of the offspring. Specific target genes include SLC6A4, NR3C1, OXTR, BDNF, and FKBP5. The central hypothesis of this project is that the exposure to the COVID-19-related prenatal maternal stress may affect infants' outcomes from birth to 12 months partially through increased methylation of target genes involved in stress regulation. The main goal is to investigate the association between Covid-19 disease in pregnancy or COVID-19-related PMS in women pregnant during the first 9 months of the year 2020 and the emotional, social, and cognitive developmental outcomes in their infants from birth to 12 months. Additionally, the role of target genes methylation in mediating this association will be investigated. Mothers and their infants will be enrolled from the delivery units of eleven neonatal facilities located in Northern Italy's COVID-19 contagion hotspot. One group will be enrolled from April to October 2020 (COVID-Exposure Pregnancy, CEP), a second group will be enrolled from April to October 2021 (Non-Exposure Pregnancy, NEP). Moreover, the CEP group will include mothers positive or exposed to COVID-19-related MPS during different trimesters of pregnancy, allowing within-group comparisons on developmentally sensitive time windows. Within 48 hours from baby delivery, saliva samples will be obtained from CEP and NEP newborns, immediately stored at -20°C and analyzed for epigenetic analyses using Next-Generation Sequencing. At 3 and 6 months, mothers will be asked to fill-in validated and reliable questionnaires on the emotional and social-behavioral development of their infants. At 12 months, infants' stress regulation and maternal sensitivity will be evaluated through video recording of mother-infant interactions. This study will provide unprecedented relevant insights on the biochemical mechanisms underlying the impact of Covid-19 disease and the related PMS on human offspring's developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Italian nationality or full mastery of Italian language to access on-line questionnaires without support
* No prenatal pathologies or perinatal risks
* Maternal age higher than 18 years
* Newborns' gestational age equal or higher than 37 weeks

Exclusion Criteria:

* Single-parent mothers
* Medically assisted conception
* Infants' genetic or metabolic comorbidities
* Perinatal injuries or sensorial deficits

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be mother-infant dyads as defined in the Eligibility Criteria section. Maternal age equal or greater than 18 years. Infants' will be enrolled at birth and followed-up to 12 month-age.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Infant negative emotionality | At 12 months of infants' age
  Measure of infant Negative Emotionality through the Infant Behavior Questionnaire - Revised questionnaire. Negative Emotionality mean score ranges from 1 to 7 and higher scores reflect higher negative emotionality.

SECONDARY OUTCOMES:
Infants' target gene methylation status | At birth
  Methylation status of the following target genes: BDNF, FKBP5, NR3C1, OXTR, SLC6A4

OTHER OUTCOMES:
Maternal target gene methylation status | At delivery
  Methylation status of the following target genes: BDNF, FKBP5, NR3C1, OXTR, SLC6A4
Maternal mental health | At 3, 6, and 12 months of infants' age
  Measure of maternal mental health obtained through the State dimension of the Stait-Trait Anxiety Inventory. The score ranges from 20 to 80, with a clinical cut-off set at 40. Higher scores reflect higher anxiety.
Maternal sensitivity | At 12 months of infants' age
  Maternal sensitivity measured by behavioral codings of mother-infant videorecorded interactions

CONTACTS AND LOCATIONS:
Overall Officials: Livio Provenzi, PhD, Principal Investigator — University of Pavia
Locations (1):
- IRCCS Mondino Foundation, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Provenzi L, Grumi S, Giorda R, Biasucci G, Bonini R, Cavallini A, Decembrino L, Drera B, Falcone R, Fazzi E, Gardella B, Giacchero R, Nacinovich R, Pisoni C, Prefumo F, Scelsa B, Sparta MV, Veggiotti P, Orcesi S, Borgatti R; MOM-COPE Study Group. Measuring the Outcomes of Maternal COVID-19-related Prenatal Exposure (MOM-COPE): study protocol for a multicentric longitudinal project. BMJ Open. 2020 Dec 31;10(12):e044585. doi: 10.1136/bmjopen-2020-044585. PMID 33384402